CLINICAL TRIAL: NCT00927381
Title: Retrospective Evaluation of Treatments and Outcomes Associated With Antivenom Therapy For Crotaline Snakebite - A Comparison Of Severe To Mild/Moderate Envenomations
Brief Title: Retrospective Evaluation of CroFab - Efficacy in Severe Envenomation
Status: Completed | Type: Observational
Sponsor: BTG International Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: MC03/03/05
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Snake Envenomation
MeSH Terms: conditions — Snake Bites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Severe envenomation: Patients with a calculated severity score of 5 or 6 were included in this group.
- Minimal/Moderate Envenomation: Severity Score less than 5

SUMMARY:
Retrospective observational review of severe envenomation treatment with CroFab

DETAILED DESCRIPTION:
The objective of this study is to use previously collected retrospective observational data to compare treatment and outcome in patients treated with CroFab who have a severe envenomation to those with a mild/moderate envenomation.

ELIGIBILITY:
Inclusion Criteria:

* Must involve treatment of a human patient with CroFab between January 1, 2002 and December 31, 2004
* The record must contain all of the following:

  1. Clinical signs/symptoms prior to the first dose of antivenom,
  2. Documentation of all doses of antivenom used to treat the patient,
  3. Indication of whether or not initial control was achieved with antivenom.

To be included in the Efficacy Evaluable Population (EEP) in the current analysis, each record must meet the following criteria:

* Must contain enough information to calculate a severity score based on the 7-point severity scale.
* All records were included in the Safety Population in the current analysis.

Exclusion Criteria:

* Any cases identified that do not meet the inclusion criteria were excluded, including cases not treated with CroFab.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients bitten by a pit viper and treated with CroFab between January 1, 2002 and December 31 2004.
Sampling Method: Non-Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2005-01; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Severity score: in order to assess response to therapy, severity scores were calculated and compared across all recorded time points. | at baseline and following treatment with CroFab

SECONDARY OUTCOMES:
The presence of venom effects, comparison of venom effects over time, initial control of venom effects, recurrence of venom effects, and delayed onset of venom effects. | following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Dart, MD, PhD, Principal Investigator — Rocky Mountain Poison and Drug Center
Locations (1):
- Rocky Mountain Poison and Drug Center, Denver, Colorado, United States